CLINICAL TRIAL: NCT06737718
Title: Use of Eye Tracking to Study Social Perception Abnormalities in Children With Angelman Syndrome
Acronym: EYEANGEL
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241267; 2024-A02021-46 (Other: ID RCB number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Angelman Syndrome
Keywords: Angelman syndrome; Eye tracking; Social perception
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Children with Angelman syndrome followed at Necker-Enfants Malades hospital, Assistance Publique-Hôpitaux de Paris in the Centre Expert Angelman.
- Controls: Healthy volunteer children from the patients' entourage, without known neurological, genetic or psychiatric pathology.

INTERVENTIONS:
Other: Eye tracking — The eye-tracking session will take place in the Pediatric Radiology department of Necker Hospital. The child will be seated in front of a computer screen. Films and images with social and/or non-social content will be shown to the children. The session will be unique, will last approximately 15 minutes and will not involve any constraints for the child.
  Eye tracking allows to measure where and how a person looks. An infrared light is emitted towards the subject's eye. It is reflected there and a camera records the reflections generated, allowing a real-time calculation of the position of the gaze. The technique is harmless and non-invasive.
Other: Data collection from patients' medical files — Data collection from patients' medical files:
  * Brain imaging data if this examination was carried out as part of the patient's care,
  * Angelman syndrome genotypes.

SUMMARY:
Angelman syndrome (AS) is a rare neurogenetic disorder that affects approximately 1 in 15,000 children - approximately 500,000 people worldwide. It is a major neurodevelopmental disorder characterized by severe developmental delay with significant intellectual disability, lack of oral language, motor, balance, and sensory impairments.

While basic research and clinical trials are progressing, the scientific community is still searching for key biomarkers to assess significant improvements in individuals participating in clinical trials.

Eye tracking has been widely used in the diagnosis of social perception abnormalities in children with autism spectrum disorder, as has already been the case for other rare neurodevelopmental diseases. However, few studies have highlighted the usefulness of eye tracking as a diagnostic tool for social behavioral disorders in individuals with Angelman syndrome. Given the prevalence of autistic-like symptoms in patients with AS, if eye-tracking can identify abnormalities in social perception in children with Angelman syndrome, these measurements could become a biomarker for therapeutic studies in these patients.

DETAILED DESCRIPTION:
Angelman syndrome (AS) is a rare neurogenetic disorder that affects approximately one in 15,000 children - approximately 500,000 people worldwide. It is a significant neurodevelopmental disorder. It is characterized by severe developmental delay with significant intellectual disability, lack of oral language, motor, balance and sensory disorders. Individuals with Angelman syndrome have specific behavioral characteristics, including happy behavior, characterized by laughter, smiling and frequent excitability.

The landscape of treatment research for Angelman syndrome has changed significantly over the past 10 years with more and more players getting involved. Different gene therapy avenues are in advanced research phases and some treatments for downstream therapies and gene activation of the paternal allele have already been in clinical trials for more than 3 years.

As basic research and clinical trials progress, the scientific community is still looking for key biomarkers to assess significant improvements in individuals participating in clinical trials.

Eye tracking has been widely used in the diagnosis of social perception abnormalities in children with autism spectrum disorder, and this has also been the case for other rare neurodevelopmental diseases. However, few studies have highlighted the usefulness of eye tracking as a diagnostic tool for social behavior disorders in individuals with Angelman syndrome.

Given the prevalence of autistic-like symptoms in patients with AS, if eye-tracking can identify social perception abnormalities in children with Angelman syndrome, these measurements could become a biomarker for therapeutic studies in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 40 children with Angelman syndrome diagnosed by genetic assessment or EEG.
* 20 healthy volunteer control children with no known genetic or psychiatric neurological pathology.
* Aged between 3 - 17 years.
* Male or female.
* Holders of parental authority and minors informed and not opposed to participation in the research.

Exclusion Criteria:

* Refusal to participate in the study.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Angelman syndrome followed at Necker-Enfants Malades hospital, Assistance Publique-Hôpitaux de Paris in the Centre Expert Angelman and healthy volunteer children from the patients' entourage, without known neurological, genetic or psychiatric pathology.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Abnormalities of social perception in children with Angelman syndrome | Time 0
  Social perception abnormalities in children with Angelman syndrome will be studied using eye tracking.
  Social perception will be measured during the eye-tracking test by the number of fixations in social and non-social regions.

SECONDARY OUTCOMES:
Description of brain abnormalities in children with Angelman syndrome | Time 0
  Description of measurements from anatomical and functional brain imaging data (radiological analysis, grey matter analysis, white matter analysis, resting cerebral blood flow analysis) available in children with Angelman syndrome participating in the study and who previously have undergone a MRI as part of their routine care.
Correlation measures between eye-tracking data and multimodal brain imaging data | Time 0
  Description of correlations of eye tracking data and multimodal brain imaging data (anatomical and functional) from children with Angelman syndrome participating in the study for whom brain imaging data has already been acquired as part of the child's routine care.
Description of potential correlations between eye-tracking data and different genotypes of Angelman syndrome | Time 0
  Investigate potential correlations measurements between eye-tracking data and different genotypes of Angelman syndrome: Deletion, Mutation, IPD, Uniparental disomy, others;
Description of potential link between eye-tracking and brain imaging data of children with Angelman syndrome to the overall eye-tracking results of children with autism spectrum disorders | Time 0
  Comparison of eye-tracking and brain imaging data obtained in children with Angelman syndrome and the same data from children with autism spectrum disorders, available in the laboratory database.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie MD, PhD Boddaert, Study Director — Assistance Publique - Hôpitaux de Paris; Monica MD Zilbovicius, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No